CLINICAL TRIAL: NCT04822129
Title: A Comparison of Two Approaches to Developing Brain Health Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Raymond Ownby, M.D., Professor and Chair, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pending
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Older Persons Interested in Improving Their Brain Health
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Intervention for TAU group: Actual participation in the intervention will begin with the first videoconference. The general format for each conference will be a brief presentation (10-15 minutes) by Dr. Ownby on a specific topic related to brain health, with the remainder of the time spent in discussion of the topic's importance and in answering participants' questions about the topic or about any other concerns they have related to developing a brain healthy lifestyle. The first videoconference will also provide participants with an overview of the daily log form, instructions for completing it and entering results every week in RedCap, and a reminder on the process of compensation for completion of the logs.
  Interventions: Behavioral: Treatment as Usual
- Cogtrastim model (Experimental): The study intervention for this group will include a review of the Cogtrastim model and explicit discussion of the possible mechanisms of action of various activities that have been shown to be associated with better health in general and, where supported by evidence, better mental functioning in older persons. Persons in this group will be encouraged to select brain health activities based on the model. Early videoconference sessions will also focus on strategies for behavior change, including realistic goal setting, problem solving about possible difficulties, and assistance in formulating a written plan to improve brain health. Participants will be encouraged to develop a written program for brain health and to also develop self-monitoring habits.
  Interventions: Behavioral: Cogtrastim Model

INTERVENTIONS:
Behavioral: Treatment as Usual — Treatment as usual will provide participants with basic information that is readily available as well as the encouragement to develop a brain health program that may be available from medical professionals.
  Other Names: TAU
  Arms: Treatment as usual
Behavioral: Cogtrastim Model — The study intervention for this group will include a review of the Cogtrastim model and explicit discussion of the possible mechanisms of action of various activities that have been shown to be associated with better health in general and, where supported by evidence, better mental functioning in older persons. Persons in this group will be encouraged to select brain health activities based on the model.
  Other Names: Cogtrastim
  Arms: Cogtrastim model

SUMMARY:
This is a research study, designed to test and create new ideas that other people can use. The purpose of this research study is to evaluate two ways of helping people learn to keep their brain healthy. Research has shown that things like exercise, diet, and computer-based cognitive training (doing things that make you think and remember on a computer or tablet) may help older persons maintain their mental functioning as they get older. We want to look at two ways for people to a develop brain healthy lifestyle that they can use and even enjoy. If we find that one of the ways of developing a brain healthy lifestyle is better than the other, other older persons may be able to use it, too. When we say "brain healthy lifestyle," we mean doing things that help to keep you healthy, like exercising and following a good diet. We also mean doing things that may help you think better and maintain your thinking and reasoning as you get older.

DETAILED DESCRIPTION:
Overview: Participants will complete a baseline battery of self-report and cognitive measures before and after 12 weeks of weekly videoconferences and diaries of brain health-related activities completed during weeks 1, 6, and 12. They will be randomly assigned to one of two groups: (1) treatment as usual (TAU), in which they will receive basic information about a brain healthy lifestyle (topics such as diet, exercise, computer-based cognitive training, meditation as well as others) and encouraged to develop a brain-health lifestyle or (2) an intervention based on the Cogtrastim model combined with behavior change support. This model posits that brain healthy lifestyle should encompass activities focused on one of three basic mechanisms related to brain health. Model-based activity choices will be integrated with an intensive behavior change intervention focused on realistic goal setting, self-monitoring, problem solving barriers to behavior change, and developing strategies for behavior maintenance.

Rationale for TAU: The intervention to be used in the treatment as usual group is a reasonable representation of what many older persons face in finding out about the importance of brain health, selecting from the broad range of potential brain health activities, and changing their health-related behaviors. A great deal of information is available online and in books. Many models of programs for brain health recommend multiple activities or interventions with little guidance on selection or prioritizing them. The TAU intervention will mirror this situation, providing participants with multiple resources from which to choose activities and methods of behavior change.

Baseline assessment: After completion of the informed consent interview and the participants have given consent to be involved in study procedures, the researchers will complete an interview with participants focused on medication use, health status, and demographic information. They will then be given links to self-report questionnaires on RedCap and sent an invitation e-mail to complete a cognitive assessment on the Cognifit website.

Measures will include the Memory Self-Efficacy Scale, Alzheimer Disease Risk Inventory (ADRI), Perceived Stress Scale, Dementia Knowledge Assessment Scale, risk subscale, PROMIS Cognitive Function, Self-Report Measure of Cognitive Abilities, Technology Use Questionnaire, and the NIH Toolbox General Life Satisfaction Questionnaire.

Cognifit assessment: This is a commercially-available product previously used in studies of computer-based cognitive training in older adults. The Cognitive Assessment Battery for People Over 55 (CAB-AG) requires 20 to 30 minutes and measures various mental abilities as well as briefly assessing mental well-being. It is a standard commercially-available product. It provides a general score as well as subscores in domains of reasoning, memory, attention, coordination, and perception.

INTERVENTIONS

Intervention for TAU group: Actual participation in the intervention will begin with the first videoconference. The general format for each conference will be a brief presentation (10-15 minutes) by a researcher on a specific topic related to brain health, with the remainder of the time spent in discussion of the topic's importance and in answering participants' questions about the topic or about any other concerns they have related to developing a brain healthy lifestyle. The first videoconference will also provide participants with an overview of the daily log form, instructions for completing it and entering results every week in RedCap, and a reminder on the process of compensation for completion of the logs.

Intervention for Cogtrastim group: The study intervention for this group will include a review of the Cogtrastim model and explicit discussion of the possible mechanisms of action of various activities that have been shown to be associated with better health in general and, where supported by evidence, better mental functioning in older persons. Persons in this group will be encouraged to select brain health activities based on the model. Early videoconference sessions will also focus on strategies for behavior change, including realistic goal setting, problem solving about possible difficulties, and assistance in formulating a written plan to improve brain health. Participants will be encouraged to develop a written program for brain health and to also develop self-monitoring habits.

All participants will be given access to the study website at www.sfbrainhealth.com which will serve as a compendium of links to relevant and reviewed brain health resources (e.g., links to material on older adults and exercise on the websites of the Centers for Disease Control and the National Institute on Aging).

All participants will be asked to complete a baseline assessment (RedCap questionnaires and Cognifit cognitive assessment) prior to participating in any other study procedures. They will be asked to complete a daily study diary of their training activities for seven days in weeks one, six, and 12 of the study. They will be given access to the Cognifit training activities after completion of the baseline assessments.

Cognifit training program: The Cognifit training program is based on an automated algorithm that selects a variety of activities based on the participant's strengths and weaknesses as well as their training history. At a summary level, Cognifit identifies which cognitive abilities (of those covered in the applied training) are most in need of improvement, and how long it has been since a cognitive ability has been trained. When, based on a series of weightings of these variables, it is decided which cognitive capacity is to be trained, the system checks which activities best train these cognitive capacities and how long it has been since they were trained. In this way, the system ensures that training focuses heavily on the cognitive abilities (and consequently on the tasks) that the user needs to train the most, but without forgetting to continue training the cognitive abilities that the user has in good condition.

Participants in both groups will be given access to weekly videoconferences brain health topics and encouraged to develop a plan to improve their brain health during the 12 weeks of the study. At the conclusion of this period, participants will be asked to complete the same battery of measures they had completed at the beginning with the addition of a questionnaire asking for ratings of the study interventions. They will be scheduled for an exit interview during which a semi-structured interview outline will be used to assess participants' reactions to the study and elicit their suggestions for improving future versions.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be community-dwelling persons 50 years of age and older who are interested in developing a more brain healthy lifestyle and are willing to participate in a 12-week study of brain health. They must have access to a stable internet connection that will allow them to communicate with the researchers by e-mail, complete online assessments and cognitive training, and participate in videoconferences.

Exclusion Criteria:

* Persons who are not community dwelling (i.e., do not live independently) as persons in a nursing facility will not be eligible, however, persons who live independently in a facility that provides a range of support will be eligible. If, in the course of the informed consent process, it appears that the person does not have the ability to provide meaningful informed consent, they will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Australian National University Alzheimer's Disease Risk Index (ANU-ADRI) | Three months
  A composite measure of personal characteristics related to risk for cognitive decline in older persons. Scores range from 0 to 76 with higher scores indicating higher exposures to risk factors for dementia.

SECONDARY OUTCOMES:
Memory Self Efficacy Scale | Three months
  A brief measure of how participants feel about their memory functioning. Scores range from 10 to 70, with higher scores indicating self-report of fewer memory problems (better memory functioning).
Dementia Knowledge Scale, Risk subscale | Three months
  A brief assessment of lifestyle factors related to risk for developing dementia. Scores range from 0 to 6, with higher scores indicating greater knowledge of risk factors for dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L Ownby, MD, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- Center for Collaborative Research, Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to qualified researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Twelve months after study completion
Access Criteria: Any researcher who presents a reasonable plan for a follow-up data analysis will be accommodated.

REFERENCES:
- [Derived] Ownby RL, Davenport R. An Online Shared Decision-making Intervention for Dementia Prevention: A Parallel-group Randomized Pilot Study. Curr Alzheimer Res. 2023;20(8):577-587. doi: 10.2174/0115672050274126231120112158. PMID 38047365
- See also: Study website with links to brain health information. — https://sfbrainhealth.com
- See also: Page on study website with study flyer and contact form. — https://sfbrainhealth.com/study